CLINICAL TRIAL: NCT02689856
Title: A Randomized, Dose-Ranging, Double Blind Study of Lidocaine Hydrochloride and/or Hydrocortisone Acetate (Alone or in Combination) in the 14-Day Twice-Daily Treatment of Grade I or II Hemorrhoids
Brief Title: Safety and Efficacy of Hydrocortisone and Lidocaine Treatment of Grade I and II Hemorrhoids
Acronym: Hydro/Lido
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Citius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 143-6151-201
Record Dates: First submitted 2016-02-17; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — hydrocortisone acetate; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Vehicle cream (Placebo Comparator): Placebo control base cream
  Interventions: Drug: Placebo control
- 3% hydrocortisone (Experimental): 3% Hydrocortisone acetate cream
  Interventions: Drug: Hydrocortisone acetate
- 0.5% hydrocortisone (Experimental): 0.5% Hydrocortisone acetate cream
  Interventions: Drug: Hydrocortisone acetate
- 5% lidocaine (Experimental): 5% Lidocaine hydrochloride cream
  Interventions: Drug: Lidocaine hydrochloride
- 1% lidocaine (Experimental): 1% Lidocaine hydrochloride cream
  Interventions: Drug: Lidocaine hydrochloride
- 3% Hydro 5% Lido (Experimental): Hydrocortisone acetate and lidocaine hydrochloride at 3% and 5% cream
  Interventions: Drug: Hydrocortisone acetate and lidocaine hydrochloride
- 0.5% Hydro 1% Lido (Experimental): Hydrocortisone acetate and lidocaine hydrochloride at 0.5% and 1% cream
  Interventions: Drug: Hydrocortisone acetate and lidocaine hydrochloride

INTERVENTIONS:
Drug: Hydrocortisone acetate and lidocaine hydrochloride — Hydrocortisone and lidocaine in combination
  Arms: 0.5% Hydro 1% Lido; 3% Hydro 5% Lido
Drug: Placebo control — Vehicle cream alone
  Arms: Vehicle cream
Drug: Hydrocortisone acetate — hydrocortisone alone
  Arms: 0.5% hydrocortisone; 3% hydrocortisone
Drug: Lidocaine hydrochloride — lidocaine alone
  Arms: 1% lidocaine; 5% lidocaine

SUMMARY:
The objectives of this study are to assess the potential contribution of lidocaine hydrochloride or hydrocortisone acetate, alone or in combination, in topical cream preparations in the treatment of Grade I or II hemorrhoids and to demonstrate the safety and efficacy of the test articles when applied twice daily for 14 days in subjects with Grade I or II hemorrhoids. These products reflect common drug combinations of lidocaine hydrochloride or hydrocortisone acetate found in many prescription hemorrhoid products.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel group comparison study in approximately 196 enrolled subjects (~28 subjects/test article) at approximately eight (8) sites. A minimum of 147 patients will be enrolled. Up to an additional 56 subjects (up to 196 subjects) may be enrolled based on enrollment rates and availability of patients. Enrollment status reports will be periodically generated, and based on enrollment experience, additional randomization blocks will be assigned to sites with the potential to enroll additional subjects over a reasonable period of time.

Male and female subjects, ages 18 years and older, with a clinical diagnosis of symptomatic Grade I or Grade II hemorrhoids will be randomized to treatment with one of seven (7) test articles (1:1 for all groups):

1. Vehicle Cream
2. 3% Hydrocortisone Acetate Cream
3. 0.5% Hydrocortisone Acetate Cream
4. 5% Lidocaine Hydrochloride Cream
5. 1% Lidocaine Hydrochloride Cream
6. 3% Hydrocortisone Acetate Cream and 5% Lidocaine Hydrochloride Cream
7. 0.5% Hydrocortisone Acetate Cream and 1% Lidocaine Hydrochloride Cream

The test articles will be applied twice daily for two (2) weeks (14 days) to the peri-rectal area as well as the distal aspect of the anal canal using the product applicator tip.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female 18 years of age or older, in generally good health. Females must be post-menopausal, surgically sterile or have a negative urine pregnancy test (UPT) at the Baseline Visit and agree to use birth control during the study.
2. Subject has provided written and verbal informed consent.
3. Subject presents to the clinic with clinically confirmed symptomatic Grade I or II hemorrhoids (GSDS ≥ 2).
4. Subject is willing and able to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

1. Subject is female and lactating or planning to become pregnant during the study.
2. Subject has anorectal condition(s) such as malignant tumors of the anus or rectum, fistula-in-ano or chronic sepsis, fissure-in-ano, incontinence, condylomata and Grade III and IV hemorrhoids.
3. Subject has a history of previous proctological surgery or has active inflammatory bowel disease.
4. Subject may use stool softeners, but shall be on a stable regimen for at least 28 days prior to enrolling in the study.
5. Subject used the following systemic, oral or topical therapies for the periods specified prior to entry into the study:

   * Within 1 day: Topicals of any kind to the rectal/peri-rectal area.
   * Within 1 week: Over the counter (OTC) or prescription treatments labeled or intended for the treatment of hemorrhoids or that could have a significant effect in the opinion of the investigator including but not limited to steroids, OTC and prescription hemorrhoid products, among others.
6. Subject has a current history of an uncorrected coagulation defect or concurrently uses anticoagulants (except aspirin or non-steroidals).
7. Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical, systemic or surgical therapy.
8. Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
9. Subject has any condition which, in the Investigator's opinion, would make it unsafe or preclude the subject's ability to fully participate in this research study.
10. Subject is unable to communicate or cooperate with the Investigator due to language problems, poor mental development, impaired cerebral function or physical limitations.
11. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
12. Subject is currently enrolled in an investigational drug or device study.
13. Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (Baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Global score of disease severity | up to 14 days
  A measure overall discomfort on a scale of 0 to 5

SECONDARY OUTCOMES:
Individual signs and symptoms | up to 14 days
  Has the subject received relief of pain, itching, bleeding or other reported symptoms evaluated on a scale of 0 to 5.
Onset of relief of symptoms | 4 hours following product administration
  How fast does the subject feel relief of symptoms measured in time after application of the drug.
Recurrence of symptoms | 4 hours following product administration
  When do the symptoms return measured in time after application of the drug.
Severity and frequency of adverse events | 14 days
  Assessment of severity and frequency of adverse events.
Laboratory assessment | 14 days
  Assessment of changes in blood chemistry, hematology and urinalysis at day 14 compared to baseline.
Electrocardiography | 14 days
  Assessment of changes in ECG parameters at day 14 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Lader, Ph.D., Study Director — Citius Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No